CLINICAL TRIAL: NCT00187525
Title: A 52 Week Open Label Trial of Memantine for Frontotemporal Lobar Degeneration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAM-02A
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Frontotemporal Lobar Degeneration
MeSH Terms: conditions — Frontotemporal Lobar Degeneration | interventions — Memantine

INTERVENTIONS:
Drug: Memantine

SUMMARY:
This is a 52-week, multicenter, open label trial of memantine (Namenda) for frontotemporal lobar degeneration (FTLD). The goal is to determine the safety and tolerability of this FDA-approved medication for Alzheimer's Disease in patients with FTLD. Secondary outcome measures include cognitive batteries, rating scales for activities of daily living and neuropsychiatric symptoms. All patients receive the FDA-approved dose of this medication for Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Neary et al. Criteria for Frontotemporal Lobar Degeneration
* Age 40 -80
* CDR < 3 or MMSE > 15
* English Speaking
* Study Partner

Exclusion Criteria:

* Concurrent use of antipsychotic drugs or acetylcholinesterase inhibitors

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-05; Primary Completion 2005-10 (Actual); Study Completion 2006-10 (Actual)

REFERENCES:
- [Derived] Boxer AL, Lipton AM, Womack K, Merrilees J, Neuhaus J, Pavlic D, Gandhi A, Red D, Martin-Cook K, Svetlik D, Miller BL. An open-label study of memantine treatment in 3 subtypes of frontotemporal lobar degeneration. Alzheimer Dis Assoc Disord. 2009 Jul-Sep;23(3):211-7. doi: 10.1097/WAD.0b013e318197852f. PMID 19812461